CLINICAL TRIAL: NCT03606551
Title: EXD-959 Esthetic Ceramic Self-ligating Orthodontic Brackets and EXD-961 Related Instruments Trial: A Multicenter Case Series Study of the Performance o the EXD-959 Ceramic Bracket System in New and Intercept Orthodontic Patients
Brief Title: EXD-959 Orthodontic Brackets and EXD-961 Related Instruments Trial
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: EM-11-050006
Record Dates: First submitted 2018-07-02; First posted 2018-07-31 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Malocclusion
Keywords: Self-ligating; Orthodontic; Esthetic
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- New Orthodontic Patients: New patient subjects who are just initiating full orthodontic treatment will have their premolars, canines, and incisors bonded with the EXD-959 Bracket System, using the related EXD-961 instruments, according to the manufacturer's IFU.
  Their remaining teeth will be bonded with the brackets of the orthodontist's choice. Three of the 5 new patients recruited may be patients that the orthodontist will choose to initiate treatment with the EXD-959 study brackets being applied to the upper teeth only. Having this option will allow the investigators to recruit subjects with deeper over-bites where their standard of care would be to apply esthetic brackets on the upper teeth and metal brackets on the lower teeth.
  Interventions: Device: EXD-959 Bracket System
- Intercept Orthodontic Patients-Progress: This group will include a minimum of three, and up to 5 patients at each study site who have moved into rectangular wires; and in whom, the orthodontist- investigator believes they will be able to evaluate rotation corrections using the EXD-959 Bracket System. For example, rotation correction of the upper central incisor which will test the width of the bracket's holding points in situations that have wide teeth and greater inter-bracket distance.
  Interventions: Device: EXD-959 Bracket System
- Intercept Orthodontic Patients-Finishing: This group will include a minimum of three, and up to 5 patients per study site who are estimated to be within 4 months of completing their orthodontic treatment; and in whom, the orthodontist-investigator believes they will be able to evaluate both torque control and debonding experiences using the EXD-959 Bracket System.
  Interventions: Device: EXD-959 Bracket System

INTERVENTIONS:
Device: EXD-959 Bracket System — EXD-959 Ceramic Self-ligating Brackets are a new type of esthetic ceramic bracket developed by 3M™ Oral Care Solutions. The brackets have a sliding door and are composed of alumina (aluminum oxide) and small amounts of related oxide compounds (glass powder) to give them a clear appearance. A nickel-titanium wire serves as part of the door mechanism and is attached to the bracket using 3M ESPE™ Scotchbond™ Universal Adhesive. The brackets are classified as a Class II medical device. A FDA 510(k) submission of EXD-959 was submitted the first quarter of 2018.

SUMMARY:
The purpose of this study is to assess the performance of the EXD-959 self-ligating ceramic bracket system using EXD 961 instruments in the treatment of orthodontic malocclusion. The information gained in this study and other studies will be used to evaluate the clinical performance of the bracket system during orthodontic treatment and to substantiate marketing claims for the bracket system, open/close instrument and de-bonding instrument.

DETAILED DESCRIPTION:
This prospective case-series study will evaluate the performance of the EXD-959 ceramic bracket system at baseline (BL), 4, and 6 months post-baseline, and at the time that each subject has their study brackets debonded (approx. 4 to 24 months). Bond failures and adverse events will be tracked throughout the entire study. A total of 78 study subjects will be enrolled in this study (30 new and 48 intercept cases). The patients will be recruited from a total of 6 participating study sites.

Self-Ligating (SL) Practitioners: The sponsor will recruit 4 orthodontist-investigators who have experience using and currently use self-ligating style orthodontic brackets.

Ligating (L) Practitioners: The sponsor will recruit 2 orthodontist-investigators who do NOT currently use self-ligating style orthodontic brackets in their practices. These will be practitioners who currently use brackets that require that either metal or elastomeric ties are used to secure the archwire into the bracket-slots.

Five new and 8 intercept subjects, who meet the inclusion/exclusion criteria and consent/assent to participate, will be enrolled at each study site (n = 13 per site).

* New patient subjects who are just initiating full orthodontic treatment will have their premolars, canines, and incisors bonded with the EXD-959 brackets, using the related EXD-961 instruments, according to the manufacturer's IFU. Their remaining teeth will be bonded with the brackets of the orthodontist's choice. Three of the 5 new patients recruited may be patients that the orthodontist will choose to initiate treatment with the EXD-959 study brackets being applied to the upper teeth only. Having this option will allow the investigators to recruit subjects with deeper over-bites where their standard of care would be to apply esthetic brackets on the upper teeth and metal brackets on the lower teeth.
* Intercept patient subjects: Eight subjects will be recruited from patients who are currently undergoing orthodontic treatment. Their existing treatment will be intercepted. They will have the brackets currently on their upper and lower premolars, canines, and incisors debonded and replaced with the EXD-959 study brackets, preferably using the related EXD-961 instruments, according the manufacturer's IFU. Three of 8 new intercept patients recruited may have treatment initiated on upper teeth only.
* In order to evaluate rotation correction, torque control, bracket and bracket- door durability, and debonding experiences two types of intercept patients will be targeted:

  * Intercept - progress: this group will include a minimum of three patients at each study site who have moved into rectangular wires; and in whom, the orthodontist- investigator believes they will be able to evaluate rotation corrections. For example, rotation correction of the upper central incisor which will test the width of the bracket's holding points in situations that have wide teeth and greater inter-bracket distance.
  * Intercept-finishing: this group will include a minimum of three patients per study site who are estimated to be within 4 months of completing their orthodontic treatment; and in whom, the orthodontist-investigator believes they will be able to evaluate both torque control and debonding experiences.

As long as they recruit a minimum of 3 subjects in each intercept category, each orthodontist-investigator can then determine the total number of subjects recruited in each of the progress- and finishing-intercept groups in order to reach a total of 8 subjects. For example, at one site they might recruit 3 progress and 5 finishing subjects, while another site might recruit 4 progress and 4 finishing subjects.

In both SL and L practitioners the EXD-959 bracket system will be used in conjunction with the archwires prescribed by the treating orthodontists according to their respective treatment philosophies.

The study patients, treating orthodontists, and orthodontic staff who interact with the study subjects, the EXD brackets, and the EXD instruments will provide feedback related to specific attributes of the product at defined time-points, using the study documents provided by the study sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to voluntarily sign the consent/assent form(s);
2. Willing and able to return to the study facility for scheduled visits and recalls;
3. Have permanent dentition including first molars, premolars, canines, and incisors erupted;
4. Teeth have sound, non-carious buccal enamel, free from white-spot lesions; and,
5. Have good oral hygiene as determined by the orthodontist/dental hygienist.

   For intercept patients only:
6. Currently have brackets on their teeth; and,
7. Have begun treatment with rectangular archwires; or, who are in their finishing stage of orthodontic treatment (i.e. they have 3 to 4 months of treatment remaining).

Exclusion Criteria:

1. Currently participating in another clinical study.
2. Difficulty being compliant with study visits, such as those planning or having extensive travel commitments or who lack transportation.
3. Have mental, emotional, or developmental disabilities.
4. Have a complex/surgical case.
5. Have a deep overbite that would result in their maxillary incisor teeth occluding with the ceramic brackets on the mandibular teeth that cannot be avoided.
6. Need essential dental care, i.e., for broken teeth, grossly carious or abscessed teeth.
7. Have dental prostheses/implants that will interfere with projected teeth movement.
8. Have known allergies to product ingredients (e.g. methacrylate resin materials, nickel, chromium).
9. Have a medical or oral condition that, in the investigator's judgement, may compromise the subject's safety or interfere with the conduct and outcome of the study.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 78 male and female subjects whose permanent teeth are erupted and who will be/are undergoing orthodontic treatment at the study offices that are participating in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Performance and functionality of the EXD-959 Bracket System and Related EXD-961 instruments in correcting dental malocclusions. | The primary time-frame will be based on the Visit 4 data (12-16-wk post-baseline).
  Validate that the EXD-959 Bracket System and Related EXD-961 instruments meet the user needs based on sponsor solicited feedback from dental professionals using, and patients wearing, these new orthodontic brackets.

SECONDARY OUTCOMES:
Orthodontists' ability to correct rotated teeth in dental patients as assessed using a questionnaire with a 7-point Likert scale | The primary time-frame will be based on the Visit 4 data (12-16-wk post-baseline).
  Orthodontist-Investigators' subjective assessment of their ability to correct or straighten rotated teeth using the study brackets.
Torque control assessed using a questionnaire with a 7-point Likert scale | The primary time-frame will be based on the Visit 4 data (12-16-wk post-baseline).
  Orthodontist-Investigators' subjective assessment of their ability to achieve the desired crown-root inclination when using the study brackets. Re: Torque Control: Clinicians will complete a 7-point Likert Scale that asks them, "How satisfied are you with your ability to achieve your desired finishing goals using the study brackets?." (Orthodontists will know the meaning of torque control as it relates to the clinicians ability to use the brackets to torque the roots of teeth into an ideal location in addition to correcting the crookedness of the tooth crowns. There is a 7-point range on the scale where: #1 = Highly Satisfied and #6 = Very Dissatisfied and #7 = Not Applicable (N/A). The lower values are the better scores as they indicate how satisfied the clinicians are with their ability to achieve their desired results using the study brackets.
Study subjects' assessment of bracket comfort assessed using a a questionnaire with a 7-point Likert scale scale | The primary time-frame will be based on the Visit 4 data (12-16-wk post-baseline).
  Study subjects' subjective assessment of how comfortable the brackets feel to them. Intercept patients will complete this questionnaire for their existing brackets. Once those brackets are removed and the study bracket are placed they will be asked to complete the same questionnaire. Re: Bracket Comfort: Subjects will complete a 7-point Likert Scale that asks them, "How comfortable do the surfaces of your new braces (brackets) feel to you? There is a 7-point range on the scale where: #1 = Very Comfortable and #7 = Very Uncomfortable. The lower values are the better scores as they indicate comfort. Paired differences between bracket type will be summarized and tested for significant differences.
Bond strength; assessed using the percent of total brackets that unintentionally debond, as captured on a bond failure tracking form. | The primary time-frame will be based on the Visit 4 data (12-16-wk post-baseline).
  Bond failure rates will be computed as a percentage of individual bracket failures relative to all the teeth bonded with brackets. In addition, a 95% confidence interval of the overall bond failure rate will be computed using the Wilson Score method.
Study subjects' assessment of bracket esthetics by using a questionnaire and a 7-point Likert scale. | The primary time-frame will be based on the Visit 4 data (12-16-wk post-baseline).
  All patient-subjects will be asked to complete a form with a 7-point Likert Scale related to how they think the brackets look on their teeth. Intercept patients will complete this questionnaire for their existing brackets. Once those brackets are removed and the study bracket are placed they will be asked to complete the same questionnaire. Re: Bracket Esthetics: Subjects will complete a 7-point Likert Scale that asks them, "How well do you think your braces blend in with your teeth? There is a 7-point range on the scale where: #1 = Very Good and #7 = Very Bad. The lower values are the better scores as they indicate good esthetics. Paired differences between bracket type will be summarized and tested for significant differences. Esthetic rating differences of more than a 2-point decrease (on a 7-point Likert scale), via the individual rating at the 12-16 week visit relative to bonding, will be deemed significant.
Bracket and door durability assessed using the percent of total brackets that break, or where the door breaks, as captured on a bracket issue tracking form. | The primary time-frame will be based on the Visit 4 data (12-16-wk post-baseline).
  Sites will record all problems with any study brackets, including any issues with the bracket doors.
Ease of Removal of study brackets when treatment is completed; assessed using a questionnaire and 7-point Likert Scale | The primary time-frame will be based on the Visit 4 data (12-16-wk post-baseline).
  Orthodontist-Investigators' and/or dental assistants' subjective assessment of how easily the brackets come off of the teeth when the patient's treatment has been completed. Re: Debondng of Brackets: Clinicians will complete a 7-point Likert Scale that asks them, "Rate the ease of debonding the study brackets." There is a 7-point range on the scale where: #1 = Very Easy and #7 = Very Difficult. The lower values are the better scores as they indicate how easy it is to remove the brackets after treatment has been completed.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Lenton, MA, CCRP, Study Director — 3M
Locations (5):
- United States (5):
  - McComb Orthodontics, Culver City, California
  - Shults Orthodontics, Wellington, Florida
  - Minnesota Orthodontics, Northfield, Minnesota
  - Alvetro Orthodontics, Sidney, Ohio
  - Simply Smiles, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No